CLINICAL TRIAL: NCT01514669
Title: Analyzing the Composition of Tears and Blood for Discovery of Novel Signatures of Aggressive Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 133719
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tear Sample collection; serum sample collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: No Tx, this is observational

SUMMARY:
The purpose of this research study is to compare profiles in the blood and tears of patients with and without prostate cancer with the goal of developing a method of separating men with aggressive and non-aggressive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 35-85 years old
2. Patients who present for the evaluation of an abnormal exam or test (elevated PSA, abnormal DRE, etc.)
3. Patients who present for the evaluation of a palpable nodule or induration on prostate exam
4. Patients who meet the requirements of Group 1, 2, or 3 of the protocol

Exclusion Criteria:

1. Patient < 35 or > 85 years of age
2. Concurrent eye infection or trauma, including active conjunctivitis
3. Abnormal production of tears (too much or too little)
4. Any other conditions the PI or staff feels will not fulfill the criteria for study entry or will place the subject in a harmful environment
5. Atypia on prostate biopsy report

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from those outpatients followed in the Winthrop P. Rockefeller Cancer Institute (located at the University of Arkansas for Medical Sciences).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Tear Sample | 1 day
  Tear sample will be taken at the initial clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Alan Diekman, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States